CLINICAL TRIAL: NCT02799264
Title: A Phase I Study Evaluating the Effect of a High Fat Meal on the Pharmacokinetics of Cabotegravir in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Effect of High Fat Meal on Cabotegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Glaxosmithkline/Quintiles (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205696
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: fasted; healthy volunteers; cabotegravir; high fat; pharmacokinetics; randomized; Phase I; two way crossover
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabotegravir 30 mg: Sequence AB (fasted followed by fed) (Experimental): There will be two administration periods with 14 days of wash out. In Period 1, eligible subjects will receive a single tablet of cabotegravir 30 mg,(micronized 500 mg core weight) orally under fasted condition with at least 10 hours of prior fast. In Period 2, eligible subjects will receive single tablet of cabotegravir 30 mg, micronized 500 mg core weight orally following a high fat meal. Blood samples will be withdrawn from subjects prior to dosing and upto 8 days after the last dose of cabotegravir.
  Interventions: Drug: Cabotegravir 30 mg
- Cabotegravir 30 mg: Sequence BA (fed followed by fasted) (Experimental): There will be two administration periods with 14 days of wash out. In Period 1, eligible subjects will receive single tablet of cabotegravir 30 mg, micronized 500 mg core weight orally following a high fat meal. In Period 2, eligible subjects will receive a single tablet of cabotegravir 30 mg, micronized 500 mg core weight orally under fasted condition with at least 10 hours of prior fast. Blood samples will be withdrawn from subjects prior to dosing and upto 8 days after the last dose of cabotegravir.
  Interventions: Drug: Cabotegravir 30 mg

INTERVENTIONS:
Drug: Cabotegravir 30 mg — Cabotegravir (GSK1265744B ) is available as white to almost white, oval shaped, film coated tablet, of weight 515 mg. The tablet contains micronized cabotegravir, lactose monohydrate, microcrystalline cellulose, hypromellose, sodium starch glycolate, and magnesium stearate. Each tablet is equivalent to 30 mg cabotegravir and needs to be taken orally with 240 mL of water. Cabotegravir tablet will be administered to subjects either in fasting condition or following a high fat meal.

SUMMARY:
Cabotegravir is being developed for the treatment of human immunodeficiency virus (HIV) 1 infection. Specifically, it is being developed as a component of a 2-drug maintenance regimen (post-induction of viral suppression) that includes rilpivirine. Rilpivirine requires food for optimal absorption; therefore the recommended intake of cabotegravir in the planned Phase 3 treatment studies is with food regardless of fat or calorie content, when administered along with rilpivirine. This is a single-center, randomized, open-label, two-way crossover study in healthy adult subjects to assess the effect of a high fat meal on the single dose pharmacokinetics of CAB 30 mg. Approximately, 24 subjects will be enrolled in the study and will be screened for 30 days. Twelve subjects with at least 10 hours of fasting will be randomized to receive a single dose of cabotegravir orally (Schedule 'A'). The remaining 12 subjects will receive a single dose of cabotegravir orally along with high fat meal (Schedule 'B'). After 15 days, the subjects earlier undergoing 'Schedule A' will be switched to 'Schedule B' and those undergoing 'Schedule B' will undergo 'Schedule A'. All the subjects will be followed up to 30 days from the day of receiving first dose of cabotegravir to evaluate the effect of a high fat meal on the pharmacokinetics of cabotegravir.

ELIGIBILITY:
Inclusion Criteria:

* An eligible subject should be between 18 to 65 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the medical monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilograms (kg) and body mass index (BMI) within the range 18.5 to 31.0 kilograms per squared meter (kg/m^2) (inclusive).
* Male or female subjects. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

  1. Non reproductive potential defined as:

     Pre menopausal females with one of the following:
     * Documented tubal ligation
     * Documented hysteroscopic tubal occlusion procedure with follow up confirmation of bilateral tubal occlusion
     * Hysterectomy
     * Documented bilateral oophorectomy
     * OR has only same sex partners, when this is her preferred and usual lifestyle Post menopausal is defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post menopausal status prior to study enrolment
  2. Reproductive potential and agrees to follow one of the options listed in the modified list of highly effective methods for avoiding pregnancy in females of reproductive potential (FRP) from 30 days prior to the first dose of the study medication and until after the last dose of the study medication and completion of the follow up visit. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception
* Capable of giving signed informed consent that includes compliance with the requirements and restrictions listed in the consent form and in the protocol
* Alanine aminotransferase (ALT), alkaline phosphatase, and bilirubin <=1.5x Upper Limit of Normal (ULN ) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of clinically significant cardiovascular disease including:

  * Exclusion criteria for screening electrocardiogram ([ECG] a single repeat is allowed for eligibility determination) showing <45 and >100 beats per minute in males and <50 and >100 beats per minute in females; >120 msec of QRS duration for both males and females; and >450 msec of QTcF interval for both males and females
  * Evidence of previous myocardial infarction (pathologic Q waves, S T segment changes [except early repolarization])
  * History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease
  * Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block (AV) block (2nd degree [Type II] or higher), Wolf Parkinson White [WPW] syndrome)
  * Sinus pauses > 3 seconds
  * Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject
  * Non sustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia
* History of inflammatory bowel disease
* History of cholecystectomy or other gastrointestinal surgery (except appendectomy more than three months prior to study)
* History of peptic ulceration or pancreatitis within the preceding 6 months of screening
* History of ongoing or clinically relevant seizure disorder within the previous 2 years, including subjects who have required treatment for seizures within this time period. A prior history of seizure, with a seizure free period of at least 2 years, off antiepileptics, may be considered for enrolment if the investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the medical monitor prior to enrolment
* Any other medical condition which, in the judgment of the investigator and medical monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject. This includes but is not limited to any pre existing condition that interferes with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drug.
* Unable to refrain from the use of prescription or non prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 milliliters (mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine containing products within 30 days prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Positive hepatitis B surface antigen (HBsAg), or a positive hepatitis B core antibody (HBcAb) with a negative hepatitis B surface antibody (HBsAb) at screening or within 3 months prior to first dose of study treatment.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of the study treatment.
* A positive pre study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90 to 140 millimeters of mercury (mmHg), or diastolic blood pressure is outside the range of 45 to 90 mmHg
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half lives or twice the duration of the biological effect of the investigational product (whichever is longer); however, the subject should not be participating in another clinical trial at the time of screening, and by the time of first dosing should not be within the time periods listed above
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve from time zero (pre dose) extrapolated to infinite time of cabotegravir | Pre dose, 0.5 hour (h), 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on Day(D) 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  AUC (0 infinity[inf]) is defined as the area under cabotegravir plasma concentration time curve from time zero (pre dose) extrapolated to infinite time.
Area under the concentration time curve from time zero (pre dose) to last time of quantifiable concentration of cabotegravir | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  AUC (0-t) is defined as area under cabotegravir plasma concentration time curve from time zero (pre dose) to the last time of quantifiable concentration.
Maximum observed plasma concentration of cabotegravir | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  Cmax is defined as the maximum observed plasma concentration of cabotegravir.
Concentration of cabotegravir at 24 hours post dose (C24) | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  C24 is defined as the plasma concentration at 24 hours after administration of cabotegravir.

SECONDARY OUTCOMES:
Plasma terminal phase half life of cabotegravir | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  Terminal elimination half life (t1/2) is defined as the duration until observation of half of the maximum concentration of cabotegravir.
Lag time before observation of cabotegravir concentration in sampled matrix | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  tlag is the observed time prior to the first quantifiable plasma concentration of cabotegravir
Time of occurrence of maximum observed plasma concentration of cabotegravir | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  tmax is defined as the time of the maximum observed plasma concentration of cabotegravir.
Percentage of area under the concentration time curve of cabotegravir from time zero extrapolated to infinite time obtained by extrapolation | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  AUC (0-inf) is defined as the area under cabotegravir plasma concentration time curve from time zero (pre dose) extrapolated to infinite time. %AUCex is percentage of AUC(0 inf) obtained by extrapolation.
Time of last measurable concentration of cabotegravir | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  tlast is defined as the time of the last observed quantifiable concentration of cabotegravir.
Apparent clearance of cabotegravir following oral dosing | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  Clearance of a drug is a measure of rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose of cabotegravir (apparent oral clearance, CL/F) is influenced by the fraction of dose absorbed.
Apparent volume of distribution of cabotegravir | Pre dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post dose on D 1, D 2, D 3, D 4, D 6, D 8 each for Period 1 and Period 2
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution of cabotegravir after oral dose (Vz/F) is influenced by the fraction absorbed.
Number of subjects with adverse events and serious adverse events | Upto approx. 68 days
  An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated), temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose can result in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/ birth defect, or any other situation related to impaired liver function.
Number of subjects with severity type | Upto approx. 68 days
  Intensity of an AE is used to rate the severity of an event. The intensities can be mild (easily tolerated), moderate (sufficiently discomforting to interfere with normal activities), or severe (prevents normal activities); however, both AEs and SAEs can be assessed as severe.
Number of subjects on concurrent medications | Upto approx. 68 days
  The number of subjects starting any other medication along with cabotegravir will be analyzed.
Number of subjects with abrnormal hematological and biochemistry laboratory parameters | Upto approx. 68 days
  Subjects will be assessed for any abnormality in hematological parameters such as platelet count, red blood cells (RBC) count, hemoglobin, hematocrit, absolute white blood cell (WBC) count, reticulocyte count, RBC distribution width, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCVC), differential WBC count including neutrophils, lymphocytes, monocytes, eosinophils, basophils and any abnormality in clinical chemistry parameters such as blood urea nitrogen (BUN), creatinine, fasting glucose, sodium, potassium, chloride, calcium, total carbon dioxide, creatine phosphokinase (CPK), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), alkaline phosphatase, total and direct Bilirubin, total protein, albumin, and uric acid. Subjects will be asked to fast for at least 4 hours prior to laboratory assessments. A single repeat will be performed.
Number of subjects with abnormal electrocardiogram | At Screening (D 30 to D1), pre dose, and 4h post dose on D1
  Duplicate ECGs will be collected with the subject in a semi supine position having rested in this position for at least 10 minutes beforehand and will be collected at Baseline (Day 1) of Period 1; however, single ECGs will be performed at all other timepoints. ECGs will be performed using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate according to Fridericia's formula (QTcF) intervals.
Number of subjects with abnormal vital signs (body temperature, systolic and diastolic blood pressure, and pulse rate) | Upto approx. 68 days
  Vital signs will be measured in semi supine position after 10 minutes rest and will include temperature, systolic and diastolic blood pressure and pulse rate. Measurements that deviate substantially from previous readings will be repeated immediately. Two blood pressure (BP) and heart rate (HR) measurements will be taken at pre dose on Day 1. The mean value recorded at pre dose will be classified as Baseline. Single BP and HR will be obtained at all other timepoints during the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Patel P, Ford SL, Lou Y, Bakshi K, Tenorio AR, Zhang Z, Pan R, Spreen W. Effect of a High-Fat Meal on the Pharmacokinetics of the HIV Integrase Inhibitor Cabotegravir. Clin Pharmacol Drug Dev. 2019 May;8(4):443-448. doi: 10.1002/cpdd.620. Epub 2018 Sep 19. PMID 30230694